CLINICAL TRIAL: NCT02667860
Title: Intra-corporeal vs Extra-corporeal Anastomosis in Laparoscopically Assisted Right Hemicolectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-AIE-2015-01
Record Dates: First submitted 2016-01-13; First posted 2016-01-29 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Pain
Keywords: intracorporeal anastomosis; laparoscopic colectomy; outcomes; length of stay; analgesia; aesthetic; extracorporeal anastomosis; laparoscopic
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intracorporeal anastomosis (Experimental): Iso or anti-peristaltic side-to-side ileo-colonic anastomosis with Echelon Endopatch and closure of the defect with running suture or another firing of Echelon Endopatch. The surgical specimen will be retrieved through a Pfannenstiel incision.
  Interventions: Procedure: Intracorporeal anastomosis.; Device: Echelon Endopatch
- Extracorporeal anastomosis (Active Comparator): A transverse incision in the right upper quadrant will be performed. An iso or anti-peristaltic side-to-side ileo-colonic anastomosis with Proximate Linear Cutter device and Proximate Rel Stapler
  Interventions: Procedure: Extracorporeal anastomosis; Device: Proximate Linear Cutter

INTERVENTIONS:
Procedure: Intracorporeal anastomosis. — Iso or anti-peristaltic side-to-side ileo-colonic anastomosis with Echelon Endopatch and closure of the defect with running suture or another firing of Echelon Endopatch. The surgical specimen will be retrieved through a Pfannenstiel incision.
  Arms: Intracorporeal anastomosis
Procedure: Extracorporeal anastomosis — A transverse incision in the right upper quadrant will be performed. An iso or anti-peristaltic side-to-side ileo-colonic anastomosis with Proximate Linear Cutter device and Proximate Stapler.
  Arms: Extracorporeal anastomosis
Device: Echelon Endopatch — Use of an Echelon Endopatch Powered Device to perform an ileocolonic side-to-side anastomosis.
  Arms: Intracorporeal anastomosis
Device: Proximate Linear Cutter — Use of a Proximate Linear Cutter device to perform a side-to-side ileo-colonic anastomosis.Use of a Proximate stapler to the closure of the defect associated with the creation of the side-to-side ileo-colonic anastomosis.
  Arms: Extracorporeal anastomosis

SUMMARY:
The creation of an intracorporeal anastomosis during right hemicolectomy is regarded as superior than the extracorporeal anastomosis in terms of recovery of peristalsis, aesthetic results, analgesia requirements and length of hospital stay. The objective of this study is to compare the postoperative results of intracorporeal versus extracorporeal anastomosis in patients undergoing laparoscopic right hemicolectomy.

DETAILED DESCRIPTION:
Laparoscopic surgery has entailed a great technical revolution in colorectal surgery, providing a better and quicker return to normal functions of the patients, associating a lower morbidity and better aesthetic results compared with traditional open surgery. This study wants to find the difference between intracorporeal and extracorporeal anastomosis.

The creation of an intracorporeal anastomosis in right hemicolectomy seems superior to extracorporeal anastomosis in terms of recovery of the normal bowel function, wound size, aesthetic results and analgesia requirements. This will entail a shorter hospital stay. Several studies have demonstrated this but all of them are retrospective non randomised.

In terms of postoperative pain, the most accepted theory is that it depends on the traction of the porto-mesenteric axis. When the intracorporeal anastomosis is performed there is no traction of this mesenteric axis while in the extracorporeal anastomosis this traction is more important in obese patients.

This traction of the mesentery, as well as being one of the main factors related with postoperative pain, is responsible of the postoperative adynamic ileus, that should have a higher incidence when the manipulation is higher.

In the patients undergoing an intracorporeal anastomosis, the assistance incision will be a suprapubic Pfannenstiel. In the patients undergoing an extracorporeal anastomosis the assistance incision will be a transverse in the right upper quadrant. It is well known that the Pfannenstiel incision has a lower incidence of superficial surgical wound infection, a lower rate of incisional hernia, a lower need of analgesics, and better aesthetic results, when compared with the incision in the right upper quadrant.

All this factors should entail a lower hospital stay in patients undergoing an intracorporeal anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* Surgical procedure with curative purpose.
* American Society of Anaesthesiologists Physical Status (ASA) I, II and III.
* Elective surgery.
* Informed consent.

Exclusion Criteria:

* Denial of informed consent.
* Advanced neoplasia.
* Urgent surgery.
* ASA IV.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-07-21 (Actual)

PRIMARY OUTCOMES:
Length of stay | 1 month
  is identified when the patient has tolerated diet and has had bowel movements and is discharged from the hospital

SECONDARY OUTCOMES:
Return to normal peristalsis | 1 week
  Physiological parameter
Size of the surgical wound | 1 month
  we measure the wound in cm
Rate of Surgical Site Infection | 1 month
  clinical wound infection or positive culture
Rate of Incisional Hernia | 1 year after discharge
  Physical exploration and CT scan (performed during the follow up)
Aesthetic result | 1 month after discharge
  Questionnaire
Postoperative pain | 1 month after discharge
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Bollo, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be available upon request to the main researcher.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All the time
Access Criteria: without

REFERENCES:
- [Derived] Bollo J, Turrado V, Rabal A, Carrillo E, Gich I, Martinez MC, Hernandez P, Targarona E. Randomized clinical trial of intracorporeal versus extracorporeal anastomosis in laparoscopic right colectomy (IEA trial). Br J Surg. 2020 Mar;107(4):364-372. doi: 10.1002/bjs.11389. Epub 2019 Dec 17. PMID 31846067
- [Derived] Bollo J, Salas P, Martinez MC, Hernandez P, Rabal A, Carrillo E, Targarona E. Intracorporeal versus extracorporeal anastomosis in right hemicolectomy assisted by laparoscopy: study protocol for a randomized controlled trial. Int J Colorectal Dis. 2018 Nov;33(11):1635-1641. doi: 10.1007/s00384-018-3157-9. Epub 2018 Sep 6. PMID 30191370